CLINICAL TRIAL: NCT06136962
Title: A Comprehensive Prospective Study on the 10-Year Outcome and Late Toxicity, Quality of Life of Reduced Volume Intensity Modulated Radiation Therapy in Nasopharyngeal Carcinoma
Brief Title: Nasopharyngeal Carcinoma Treated With Reduced Volume Intensity Modulated Radiation Therapy:10-Year Outcome and Late Toxicity, Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NPC011
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a type of head and neck cancer. The last three decades of research in head and neck radiation oncology have largely focused on improvements in survival, which have mostly come at the cost of long term toxicity for surviving patients.This is an observational study that is being done to evaluate the long-term efficacy, learn about the toxicity and quality of life that survivors of nasopharyngeal carcinoma may have following treated with reduced volume intensity modulated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment with Reduced Volume Intensity Modulated Radiation Therapy
* Age 18 or above, upper limit 65
* Ability to comply with the protocol

Exclusion Criteria:

* History of recurrent nasopharyngeal disease
* A history of any physical, psychological or social condition which would impair with the ability of the patient to cooperate in this study
* Unable to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically diagnosed non-metastatic Nasopharyngeal carcinoma (NPC) patients who were treated with Reduced Volume Intensity Modulated Radiation Therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Overall survival is calculated from diagnosis to death from any cause

SECONDARY OUTCOMES:
Loco-regional failure-free survival | 10 years
  Loco-regional failure-free survival is calculated from diagnosis to the first loco-regional failure
Failure-free survival | 10 years
  Failure-free survival rate is calculated from the date of diagnosis to the date of treatment failure or death from any cause, whichever is first
Distant failure-free survival | 10 years
  Distant failure-free survival is calculated from diagnosis to the first remote failure
Quality of Life Questionnaires QLQ-C30 | 1year
  Quality of life as measured by QLQ-C30
Quality of Life Questionnaires | 1year
  Quality of life as measured by QLQ H&N35
Evaluation of late toxicities | 1year
  Clinical toxicities will be grade according to RTOG/CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No